CLINICAL TRIAL: NCT04478370
Title: Characterizing the Humoral Immune Response Against Salivary Antigens of Southeast Asian Mosquito Vectors of Malaria and Dengue With a Human Challenge Model
Brief Title: Characterizing Humoral Immune Response to Mosquito Bites
Acronym: SG6
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: National Health and Medical Research Council, Australia (Other); Burnet Institute (Other); Agency for Science, Technology and Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MAL19009
Record Dates: First submitted 2020-06-29; First posted 2020-07-20 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-08

CONDITIONS: Malaria; Dengue
Keywords: Mosquito bites; Biomarkers; Malaria vectors; Dengue vectors
MeSH Terms: conditions — Malaria; Dengue

STUDY DESIGN:
Intervention Model Description: This study is a human challenge model with five arms corresponding to controlled exposure to bites of uninfected laboratory-adapted colonies of Anopheles minimus, An. maculatus, An. dirus, Aedes. aegypti or Ae. albopictus.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- An. minimus (Experimental): This arm will be divided into 2 groups; the low-exposure groups and the high-exposure group.
  In the low-exposure group, participants will be exposed to 5 mosquito bites at weekly intervals from day 14 to day 56 (seven challenges with 5 mosquito bites/challenge over six weeks, yielding a total of 35 mosquito bites).
  In the high-exposure group, participants will be exposed to 5 mosquito bites on day 14 and then to 50 mosquito bites at weekly intervals from day 21 to day 56 (one challenge with 5 mosquito bites and six challenges with 50 mosquito bites/challenge over 6 weeks, yielding a total of 305 mosquito bites).
  Interventions: Biological: Mosquito bites
- An. maculatus (Experimental): Same as above
  Interventions: Biological: Mosquito bites
- An. dirus (Experimental): Same as above
  Interventions: Biological: Mosquito bites
- Ae. aegypti (Experimental): Same as above
  Interventions: Biological: Mosquito bites
- Ae. albopictus (Experimental): Same as above
  Interventions: Biological: Mosquito bites

INTERVENTIONS:
Biological: Mosquito bites — Participants will be exposed to mosquito bites.
  For the low-dose challenge, five 5 to 7-day-old nulliparous female imagoes (i.e. that have never blood fed before) will be introduced individual into 50 mL plastic tube covered with netting material.
  For high-dose challenge, 47 mosquitoes will be split into four plastic cups of 10 cm in diameter covered with netting material (three cups with 12 mosquitoes and one cup with 11 mosquitoes), and 3 mosquitoes will be introduced individually into 50 mL plastic tubes.
  Mosquito bites administered on participant's arm will be used to assess immediate and delayed skin reactions. Immediate and delayed skin reactions will be recorded respectively 20-30 min and 24-36 hours after the day 14 and day 21 challenges, requiring additional visits at day 15 and 22.

SUMMARY:
The characteristics of the humoral response directed against mosquito saliva antigens are not known precisely. This is a major limitation for using immunological markers as an outcome in epidemiological trials and as an indicator for operational deployment of interventions. Recent advances in the assembly of the genome of some Anopheles and Aedes mosquito vector species has facilitated the identification of new candidate peptides in silico, using the sequences of orthologous salivary gland proteins and B-cell prediction algorithms. The objective of this study is to assess the humoral immune response directed against candidate peptides following controlled exposure to laboratory-adapted colonies of An. minimus, An. maculatus and An. dirus, Ae. aegypti and Ae. albopictus.

This research will provide essential information to identify and validate immunological markers of human exposure to malaria and dengue mosquito vectors in Southeast Asia. Immunological markers would be useful to understand transmission dynamics and predict the risk of transmission as part of a surveillance system, and to assess the efficacy of vector-control interventions in entomological trials or during operational deployment of interventions in the region.

DETAILED DESCRIPTION:
This study is a human challenge model with five arms corresponding to controlled exposure to bites of uninfected laboratory-adapted colonies of Anopheles minimus, An. maculatus, An. dirus, Aedes. aegypti or Ae. albopictus. Following screening and eligibility assessment, 150 participants will be enrolled in the study using a block-randomized design stratified on the mosquito species and number of bites (35 or 305 bites in total) such as to constitute 10 groups of 15 individuals for each of the study condition. Participants will be in the study for 112 days. The baseline will consist of 2 visits over 2 weeks (day 0 and day 7).

In the low-exposure groups, participants will be exposed to 5 mosquito bites at weekly intervals from day 14 to day 56 (seven challenges with 5 mosquito bites/challenge over six weeks, yielding a total of 35 mosquito bites). In the high-exposure group, participants will be exposed to 5 mosquito bites on day 14 and then to 50 mosquito bites at weekly intervals from day 21 to day 56 (one challenge with 5 mosquito bites and six challenges with 50 mosquito bites/challenge over 6 weeks, yielding a total of 305 mosquito bites).

The number of bites and modalities of the follow up used in this study were chosen based on previous entomological investigation conducted in this area, published reports of human challenge with mosquito bites and current knowledge on the characteristic of the humoral response against saliva antigens. Both immediate and delayed skin reactions will be recorded after day 14 and day 21 challenges, requiring additional visits at day 15 and day 22. Participants with hypersensitivity to mosquito bites will be withdrawn from the study. Both capillary and venous blood samples will be collected weekly from each study participant. Eighteen venous blood samples will be collected including one sample of 2 mL drawn during screening visit, 14 samples of 8.6 mL during visits 2, 3, 6, 8, 9, 10, 11, 12, 14, 15, 16, 17, 18 and 19, and 3 samples of 18.6 mL during visits 4, 13 and 20 (178.2 mL of venous blood per participant in total). Seventeen dry blood spot (DBS) samples will be made from of 300 μL of capillary blood collected during visits 2, 3, 4, 6, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19 and 20 (5.1 mL of capillary blood per participant in total).

Candidate peptides will be identified in silico using publicly available genomes sequences and B-cell epitope prediction algorithms. The kinetic of antibody titers against candidate biomarkers will be assessed by enzyme-linked immunosorbent assay (ELISA) and mesoscale screening performed with serum and DBS specimens. Briefly, the positivity threshold of the assay will be determined using reference sera specimens from individuals not exposed to mosquito bites, as described previously. The ELISA signal measured in 60 reference sera obtained from unexposed individuals (30 Thai sera obtained from the Thai Red Cross and 30 Australian sera obtained from the Burnet Institute) will be used to define the positivity threshold of the assay. The positivity threshold of the assay will be defined as three standard deviation (SD) above the mean optic density (ΔOD) measured for the unexposed control population. A test in the study population with a ΔOD above this cut-off will be considered positive (i.e. an immune response). The specific antibody titer of study samples will be determined by performing serial dilution experiments. Serial dilution will be made from study samples and the ΔOD will be determined for each dilution. The antibody titer will be defined as the highest dilution giving a positive signal. Results obtained with DBS and serum specimens will be compared in order to assess the feasibility of using DBS samples to monitor exposure to bites of mosquitoes during epidemiological studies. Serum specimens collected during visits 4 (baseline), 13 (early after the end of exposure) and 20 (post-exposure) will also be analysed with immuno-proteomic approach (2D gel electrophoresis of salivary gland protein extracts, Western blot and mass spectrometry) yielding additional information on the antigenic properties of mosquito salivary gland proteome.

Planned Sample Size: 150 participants followed-up for 16 weeks

Participant Identification:

Study participants are defined as healthy participants aged between 18 and 60 years old and willing to participate in the study. This study will take place at the Shoklo Malaria Research Unit (SMRU) research centre in Mae Sot.

This study was funded by the Wellcome Trust under the core funding (#220211).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female participant judged by a responsible physician with no abnormality identified on a medical evaluation;
* Thai, Burmese or Karen ethnicity;
* Aged ≥ 18 to <60 years old;
* Living in Mae Sot city for the last 12 months;
* Willing to participate in the activity and able to give informed consent for participating in the study;
* Able to tolerate direct mosquito exposure.

Exclusion Criteria:

* History of travel in a malaria endemic are (rural village) in the last 12 months, or plan to do so during the study;
* Medication or condition deemed to interfere with the outcome measure by a responsible physician;
* Moderate and severe anemia (haemoglobin concentration less than 110 g/L of blood);
* Hypersensitivity or anaphylaxis to mosquito bites;
* Pregnant women

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 147 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2025-07-23 (Actual); Study Completion 2025-07-23 (Actual)

PRIMARY OUTCOMES:
Levels of specific antibody titers against candidate peptides before and during repeated exposure to laboratory-reared mosquito bites determined by ELISA and mesoscale screening. | baseline through day 112
Kinetics of specific antibody titers against candidate peptides before and during repeated exposure to laboratory-reared mosquito bites determined by ELISA and mesoscale screening. | baseline through day 112
Sequence of saliva antigens determined with an immuno-proteomic method (2D gel electrophoresis of salivary gland protein extracts, Western blot and mass spectrometry). | Day 14 through day 112

SECONDARY OUTCOMES:
Comparison of the antibody titers determined in subgroups corresponding to different level of exposure. | Day 0, 7 (baseline), 14, 21, 28, 35, 42, 49, 56 (exposure period), 63, 70, 77, 84, 91, 98, 105 and 112 (post-exposure period).
Comparison of the antibody titers determined in DBS and venous blood samples. | Day 0, 7 (baseline), 14, 21, 28, 35, 42, 49, 56 (exposure period), 63, 70, 77, 84, 91, 98, 105 and 112 (post-exposure period).

CONTACTS AND LOCATIONS:
Overall Officials: François Nosten, Principal Investigator — Shoklo Malaria Research Unit
Locations (1):
- Shoklo Malaria Research unit (SMRU), Mae Sot, Changwat Tak, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sawasdichai S, Chaumeau V, Kearney E, Wasisakun P, Simpson JA, Price DJ, Chotirat S, Renia L, Bergmann-Leitner E, Fowkes F, Nosten F. Characterizing antibody responses to mosquito salivary antigens of the Southeast Asian vectors of malaria and dengue with a human challenge model of controlled exposure: a protocol. Wellcome Open Res. 2023 Jul 11;8:135. doi: 10.12688/wellcomeopenres.19049.2. eCollection 2023. PMID 37456919

DOCUMENTS (2):
  • Study Protocol (2020-06-14): https://cdn.clinicaltrials.gov/large-docs/70/NCT04478370/Prot_001.pdf
  • Statistical Analysis Plan (2023-03-23): https://cdn.clinicaltrials.gov/large-docs/70/NCT04478370/SAP_002.pdf